CLINICAL TRIAL: NCT02806141
Title: Aerosolized Plus Intravenous Colistin Compared With Intravenous Colistin for Adjunctive Treatment of Ventilator-associated Pneumonia Due to Pandrugs-resistant Acinetobacter Baumannii in the Neonates: Randomized Controlled Trial
Brief Title: Aerosolized Plus Intravenous vs. Intravenous Colistin for VAP Due to Pandrugs-resistant A. Baumannii in Neonates
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No patient included at target sample sizes
Sponsor: Hat Yai Medical Education Center (Other)
Responsible Party: Principal Investigator, Dr. Narongsak Nakwan, Head of Division of Neonatalogy, Department of Pediatrics, Hat Yai Hospital, Hat Yai Medical Education Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HatYaiMec-Neonate
Record Dates: First submitted 2016-06-08; First posted 2016-06-20 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Pneumonia, Ventilator-Associated; Colistin Adverse Reaction; Infection Due to Multidrug Resistant Acinetobacter; Infection Resistant to Multiple Drugs
Keywords: Aerosolized colistin; Intravenous colistin
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — colistinmethanesulfonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerosolized plus intravenous colistin (Experimental): Neonates with VAP due to PDR-A. baumannii who receive aerosolized colistin (4 mg/kg/dose twice daily) plus intravenous colistin (3.5 mg/kg/dose twice daily)
  Interventions: Drug: Aerosolized plus intravenous colistin
- Intravenous colistin (Active Comparator): Neonates with VAP due to PDR-A. baumannii who receive only intravenous colistin (3.5 mg/kg/dose twice daily)
  Interventions: Drug: Intravenous colistin

INTERVENTIONS:
Drug: Aerosolized plus intravenous colistin — Aerosolized colistin at the dose of 4 mg colistin base activity (CBA)/kg twice daily (8 mg/kg/day) plus intravenous colistin at a dose of 3.5 mg CBA/kg/dose twice daily (7 mg/kg/day)
  Other Names: colistimethate sodium
  Arms: Aerosolized plus intravenous colistin
Drug: Intravenous colistin — Intravenous colistin at a dose of 3.5 mg CBA/kg/dose twice daily (7 mg/kg/day)
  Other Names: colistimethate sodium
  Arms: Intravenous colistin

SUMMARY:
This study is planned to compare the clinical efficacy and safety of aerosolized plus intravenous colistin vs. intravenous colistin as adjunctive therapy for the treatment of ventilator-associated pneumonia (VAP) due to pandrugs-resistant (PDR) Acinetobacter baumannii in the neonates.

DETAILED DESCRIPTION:
This study will evaluate the neonates with VAP due to PDR-Acinetobacter baumannii who receive aerosolized plus intravenous colistin compare with intravenous colistin as adjunctive therapy. The efficacy and safety after study will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Neonates who are admitted to the neonatal intensive care unit, Hat Yai Hospital during the study period.
* Neonates who were complicated with VAP due to PDR-Acinetobacter baumannii susceptible to colistin (by minimal inhibitory concentration (MIC) < 2 mcg/dL).

Exclusion Criteria:

* Neonates who have a major anomaly or chromosomal abnormality.
* Neonates who receive colistin prior 7 days prior to study.
* Neonates who have a significant renal dysfunction defined as a serum creatinine (SCr) >1.5 mg/dL or a decrease in urine output to < 1 mL/kg/h;

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 204 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of Patients With Cure | Through study completion, an average of 2 weeks
  Clinical outcome is classified in 4 categories: Cure, Improved, Failure, and Death
Number of Patients With Improved | Through study completion, an average of 2 weeks
  Clinical outcome is classified in 4 categories: Cure, Improved, Failure, and Death
Number of Patients With Failure | Through study completion, an average of 2 weeks
  Clinical outcome is classified in 4 categories: Cure, Improved, Failure, and Death
Number of Patients With Death | Through study completion, an average of 2 weeks
  Clinical outcome is classified in 4 categories: Cure, Improved, Failure, and Death

SECONDARY OUTCOMES:
Number of Patients With Eradication | Through study completion, an average of 2 weeks
  Microbiological response is classified in 3 categories: Eradication Persistence, Superinfection
Number of Patients With Persistence | Through study completion, an average of 2 weeks
  Microbiological response is classified in 3 categories: Eradication Persistence, Superinfection
Number of Patients With Superinfection | Through study completion, an average of 2 weeks
  Microbiological response is classified in 3 categories: Eradication Persistence, Superinfection
Number of Patients With Adverse Events That Are Related to Study Drug | Through study completion, an average of 4 weeks
  Number of Patients With Adverse Events That Are Related to Study Drug, Graded According to NCI CTCAE Version 3.0 focus on neurology, pulmonology, nephrology and metabolic/laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Narongsak Nakwan, MD, Principal Investigator — Hat Yai Medical Education Center
Locations (1):
- Narongsak Nakwan, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakwan N, Wannaro J, Thongmak T, Pornladnum P, Saksawad R, Nakwan N, Chokephaibulkit K. Safety in treatment of ventilator-associated pneumonia due to extensive drug-resistant Acinetobacter baumannii with aerosolized colistin in neonates: a preliminary report. Pediatr Pulmonol. 2011 Jan;46(1):60-6. doi: 10.1002/ppul.21324. Epub 2010 Sep 1. PMID 20812247
- [Background] Nakwan N, Lertpichaluk P, Chokephaibulkit K, Villani P, Regazzi M, Imberti R. Pulmonary and Systemic Pharmacokinetics of Colistin Following a Single Dose of Nebulized Colistimethate in Mechanically Ventilated Neonates. Pediatr Infect Dis J. 2015 Sep;34(9):961-3. doi: 10.1097/INF.0000000000000775. PMID 26065861
- [Background] Nakwan N, Usaha S, Chokephaibulkit K, Villani P, Regazzi M, Imberti R. Pharmacokinetics of Colistin Following a Single Dose of Intravenous Colistimethate Sodium in Critically Ill Neonates. Pediatr Infect Dis J. 2016 Nov;35(11):1211-1214. doi: 10.1097/INF.0000000000001263. PMID 27276179